CLINICAL TRIAL: NCT02201914
Title: Clomiphene Citrate Plus Gonadotropins and GnRH Antagonist Versus Flexible GnRH Antagonist Protocol Versus Microdose GnRH Agonist Protocol in Poor Responders Undergoing IVF: a Randomized Study
Brief Title: Clomiphene Citrate Plus Gonadotropins and GnRH Antagonist Versus Flexible GnRH Antagonist Protocol Versus Microdose GnRH Agonist Protocol in Poor Responders Undergoing IVF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bioroma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRM003
Record Dates: First submitted 2014-07-22; First posted 2014-07-28 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Poor Responders; IVF; Clomiphene Citrate; GnRH Agonist; GnRH Antagonist
MeSH Terms: interventions — Clomiphene; cetrorelix; Triptorelin Pamoate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Clomiphene citrate (Experimental)
  Interventions: Drug: Clomiphene citrate
- Daily FSH and LH plus Cetrorelix (Experimental)
  Interventions: Drug: Daily FSH and LH plus Cetrorelix
- Triptorelin plus daily FSH and LH (Experimental)
  Interventions: Drug: Triptorelin plus daily FSH anh LH

INTERVENTIONS:
Drug: Clomiphene citrate — patients receive clomiphene citrate 100 mg daily starting on day 2 for 5 days and 450 IU recombinant FSH and 225 IU recombinant LH daily starting on day 5; Cetrorelix 0,25 mg was administered daily when one or more follicle reached 13-14 mm in diameter until the hCG injection
  Arms: Clomiphene citrate
Drug: Daily FSH and LH plus Cetrorelix — Women receive an initial daily dose of 450 IU recombinant FSH and 225 IU recombinant LH starting on day 3; Cetrorelix 0,25 mg was administered daily when one or more follicle reached 13-14 mm in diameter until the hCG injection.
  Arms: Daily FSH and LH plus Cetrorelix
Drug: Triptorelin plus daily FSH anh LH — women receive short-acting Triptorelin 0,05 mg daily starting on day 1 until the hCG injection and 450 IU recombinant FSH and 225 IU recombinant LH daily starting on day 2.
  Arms: Triptorelin plus daily FSH and LH

SUMMARY:
Poor ovarian response to stimulation in IVF cycles is a challenging and frustrating condition, due to its poor prognosis in terms of chances of pregnancy and live births. Various ovarian stimulation regimens have been tried to overcome these obstacles. A simple approach is increase the dose of the gonadotropin administration, but the results in terms of pregnancy rate are very low Another commonly used stimulation regimen is the microdose GnRH agonist protocol, which takes advantage of the initial rise in endogenous gonadotropins that follows the agonist administration in the early follicular phase and subsequently prevents a premature LH surge, with fewer cycle cancellations. However, their application in poor responders, even if in small doses and for a limited period, has been questioned as they may cause oversuppression of ovarian function, leading to a prolonged cycle and increased treatment costs without improving the outcomes.

Recently, GnRH antagonists were introduced in ART treatment. They are effective in preventing a premature LH surge and allow for a more natural recruitment of follicles in the follicular phase in a non-suppressed ovary, offering a potential alternative in the treatment of these patients. However, randomized studies evaluating the efficacy of this regimen in poor responders did not show any improvements in pregnancy rates. Current approach have included the addition of oral agents such us clomiphene citrate (CC) to gonadotropins. Some authors have investigated the role of CC in addition to low dose of gonadotropins in mild stimulation regimen, demonstrating that, despite a small number of retrieved oocytes, good quality embryos were produced with a subsequent improvement in the fertilization rate, clinical pregnancy rate and live birth rate. The only study that evaluate the efficacy of CC in addition to high doses of gonadotropins in poor responders showed improving in number of retrieved oocytes, transferred embryos and biochemical pregnancy; however, clinical pregnancy rate and live birth rate remained low and showed no measurable increase.

The aim of this study was to compare the efficacy of the CC as an adjunctive to a high dose of gonadotropins in cycles with antagonist protocols with the microdose GnRH agonist and flexible antagonist protocols in women who responded poorly to ovarian stimulation, to determine whether this protocol may improve IVF outcomes, offering a valid alternative in poor responder patients treatment.

ELIGIBILITY:
Inclusion Criteria:

* poor responders in a previous IVF cycle at least 3 months before at our center and undergoing a new IVF attempt with at least two of the following criteria : I) age > 40 years old; II) basal follicular stimulation hormone (FSH) > 12 mIU/ml; III) three or fewer oocytes retrieved in the previous IVF cycle; IV) low estradiol levels on the day of human chorionic gonadotropin (hCG) administration (< 1500 pmol/ml).

Exclusion Criteria:

* body mass index > 30
* biochemical and ultrasound evidence of polycystic ovary syndrome
* stage III-IV endometriosis
* inflammatory or autoimmune disorders
* metabolic disease
* infertility medications within the past two months

Ages: 25 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-10 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | Time Frame: until 12th gestational week

SECONDARY OUTCOMES:
implantation rate | Time Frame: until 12th gestational week

CONTACTS AND LOCATIONS:
Locations (1):
- Bioroma, Rome, Rome, Italy